CLINICAL TRIAL: NCT00675311
Title: A Randomized Study of the Clinical and Economic Impact of Remote Monitoring Program With Disease Management Compared to Conventional Diabetes Disease Management Interventions
Brief Title: Remote Monitoring in Diabetes Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: Cheryl Pegus, M.D., SymCare Personalized Health Solutions, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7021
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Remote monitoring; Type 1 Diabetes; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DM-Standard (Active Comparator): The conventional disease management group will receive management under the site's usual program offering, which includes, but is not limited to, compliance with the prescribed treatment regimens, dietary management, exercise programs, and other measures recommended by the American Diabetes Association (ADA) and the Association of American Endocrinologists (AACE).
  Interventions: Behavioral: DM-Standard
- DM-Plus (Active Comparator): Plus is one of the randomized arms of the study. Patients assigned to this arm receive support from Disease Management nurses and technology that includes mobile phone client software with web-based companion software, Bluetooth glucose meter cradle, and web-based clinical management software for the clinical management team. The core of the system is the patient's cell phone which is used as an input device and which enables patients to maintain an electronic diary of information such as meal times, blood glucose, insulin use, weight, blood pressure, and exercise. The device is customizable to collect only the information relevant to the patient with diabetes and their healthcare provider. The patient with diabetes enters diary information on his or her mobile phone. No immediate or real-time information is provided to patients as part of this study.
  Interventions: Behavioral: Disease Management Plus

INTERVENTIONS:
Behavioral: DM-Standard — Device/t+ Medical Diabetes Management System
  Arms: DM-Standard
Behavioral: Disease Management Plus — Plus is one of the randomized arms of the study. Patients assigned to this arm receive support from Disease Management nurses and technology.
  Arms: DM-Plus

SUMMARY:
The primary objective of this study is to determine whether remote monitoring in diabetes management is more effective at helping patients manage their disease than a standard disease management program.

DETAILED DESCRIPTION:
To determine whether remote monitoring in diabetes management is more effective at helping patients manage their disease.

ELIGIBILITY:
Inclusion Criteria

* Between 18 and 64 years of age as of January 1, 2008
* Diagnosis of diabetes mellitus (listed ICD-9-CM diagnosis code on two or more outpatient claims, or on one or more inpatient admissions or emergency room claims in the most recent 12-month period)
* Continuously enrolled in a health plan with pharmacy and medical benefits for the most recent 12-month period or with one period of non-enrollment up to only 30 days
* Able to provide written informed consent for study participation

Exclusion Criteria

* Advanced renal disease (one or more claims in the most recent 12-month period) as defined by a claim for nephropathy or creatinine greater than 2.5 mg/dl
* Selected cancers (one or more claims in the most recent 12-month period)
* HIV/AIDS (one or more claims in the most recent 12-month period)
* Heart, liver, kidney, or multiple organ transplant (one or more claims in the most recent 12-month period)
* Cirrhosis of the liver (one or more claims in the most recent 12-month period)
* Current participation in another LifeScan study or other diabetes-related clinical trials
* Medicare is primary source of insurance coverage
* Unable to understand written and spoken English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary study measures for this study include glycemic control and LDL levels, satisfaction with diabetes care, and adherence to diabetes medications and self-monitoring recommendations | 1 Year

SECONDARY OUTCOMES:
Secondary measures include diabetes-related health-care utilization and physiologic data. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Donald Fetterolf, MD, Principal Investigator — Matria Healthcare
Locations (1):
- Marietta, Georgia, United States